CLINICAL TRIAL: NCT01670799
Title: A Pilot Trial to Study the Availability and Effect of Post-OP IV Ketorolac on Ovarian, Fallopian Tube or Primary Peritoneal Cancer, Cells Retrieved From the Peritoneal Cavity
Brief Title: Availability & Effect of Post-OP Ketorolac on Ovarian, Fallopian Tube or Primary Peritoneal Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INST 1115; NCI-2012-00917 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-08-17; First posted 2012-08-22 (Estimated); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer
Keywords: Ketorolac; Bioavailability; Pain
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms; Pain | interventions — Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketorolac (Experimental): All patients will receive a single dose of IV ketorolac for pain management for the indication of post-operative pain control. Patients less than 65 years of age and in otherwise good health will receive a 30mg IV single dose. Patients 65 years of age or greater, or who have mild renal insufficiency or are of low weight (as per section 3.2) will receive a single 15 mg dose IV ketorolac.
  In patients who have a clinical pain response and have no contraindications to multi-dose (every 6 hours over 24 hours), additional doses will be given per physician discretion based on clinical indication. Patients receiving 24 hour dosing will be eligible for sample time points after 24 hour dosing.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — This is a pilot (feasibility) trial to determine the availability, concentration and racemic mixture of a clinically indicated pain medication, ketorolac, in the peritoneal cavity and the subsequent effect on free floating ovarian cancer cells in patients after cytoreductive surgery for ovarian cancer.
  Other Names: Ketorolac tromethamine

SUMMARY:
The purpose of this study is to evaluate the anti-cancer effect of a pain medication called ketorolac (Toradol) on ovarian cancer cells in the abdominal (peritoneal) cavity after surgery for ovarian, fallopian tube or primary peritoneal cancer.

DETAILED DESCRIPTION:
Ovarian cancer is the sixth most common cancer and the seventh most common cause of cancer deaths in women across the globe. The majority of women, nearly 70%, will present with advanced stage disease that heralds a poor prognosis.

Despite aggressive treatment that still favors initial debulking surgery followed by a platinum and taxane based chemotherapy regimen, most patients relapse after achieving a complete clinical response.

Our group has shown that the ketorolac can inhibit gene activity which inhibits cell proliferation and migration.Ketorolac will be used in this study with the goal of producing specific inhibition of cell adhesion and migration in ovarian cancer cells retrieved within the peritoneal cavity after cytoreductive surgery.

ELIGIBILITY:
Inclusion Criteria:

(PRE-OPERATIVE [OP])

* Patients must be suspected of having a diagnosis of ovarian, fallopian tube or primary peritoneal cancer with a planned cytoreductive surgery
* Borderline ovarian cancer with ascites
* Eastern Cooperative Oncology Group (ECOG)/Zubrod/ Southwest Oncology Group (SWOG) performance status < 2 (Karnofsky performance status >= 70%)
* Ability to provide informed consent
* Absolute neutrophil count > 1000/uL
* Platelet count > 100'000/uL
* Serum creatinine =< 1.5 x upper limit of normal (ULN)
* Bilirubin =< 1.5 x normal
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamic pyruvic transaminase (SGPT) (alanine aminotransferase [ALT]) levels =< 2 x ULN
* No known bleeding disorders
* No known sensitivity to nonsteroidal anti-inflammatory drugs (NSAIDs)
* No active peptic ulcer disease
* No active bleeding
* SECONDARY ELIGIBILITY
* Histologic diagnosis of epithelial ovarian, fallopian tube or primary peritoneal cancer on frozen section diagnosis
* Placement of an intraperitoneal port at the time of surgery for anticipated use for adjuvant chemotherapy or management of post-operative ascites
* If epidural catheter was used - the catheter must be removed prior to treatment
* No active bleeding

Exclusion Criteria:

* Non-epithelial ovarian cancer or metastatic cancer to the ovaries
* Borderline ovarian cancer without ascites
* Presumed early stage ovarian cancer
* No clinical indication for a peritoneal port
* Active use of an epidural catheter
* Uncontrolled or unstable medical conditions
* Off study use of ketorolac or other NSAIDs prior to study administration
* Active bleeding or high risk of bleeding
* Active therapeutic anticoagulation
* Known hypersensitivity to NSAIDs
* Chronic or acute renal insufficiency as defined by a preoperative serum creatinine greater than 1.5mg/dL or creatinine clearance of < 60 ml/min
* Any co-morbid condition that' in the view of the attending physician' renders the patient at high risk from treatment complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measure levels of Ketorolac in peritoneal cavity | 24 hours
  To determine the concentration of measurable levels of R and S- Ketorolac (and the percent racemic mixture) in the peritoneal cavity after intravenous (IV) administration in the post-operative patient after cytoreductive surgery.

SECONDARY OUTCOMES:
Measure effect of IV Ketorolac on ovarian cancer cell adhesion and migration | Up to 48 hours
  The secondary endpoint of this study is to determine the effect of IV ketorolac on cell adhesion and migration of ovarian cancer cells retrieved from the peritoneal cavity after cytoreductive surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Muller, MD, Principal Investigator — UNM Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States

REFERENCES:
- See also: UNM Cancer Center website — http://cancer.unm.edu
- See also: New Mexico Cancer Care Alliance website — http://www.nmcca.org

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-01-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT01670799/Prot_SAP_000.pdf